CLINICAL TRIAL: NCT00197795
Title: Immunogenicity and Reactogenicity of a Meningococcal B Outer Membrane Vesicle Vaccine Given in a 0,6,12 Month Schedule to Health UK Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Principal Investigator, Prof. Elizabeth Miller, Consultant epidemiologist, Public Health England
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MNB1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Neisseria Meningitidis

INTERVENTIONS:
Biological: Meningococcal outer membrane vesicle vaccine "MenBVac"

SUMMARY:
To measure the serum bactericidal antibody levels and cell mediated immune responses before and six weeks after each dose of meningococcal outer membrane vesicle vaccine given at 0,6 and 12 weeks to healthy UK adults.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent given for three immunizations with MenBVac and five blood tests
* Between the ages of 18 and 55 years inclusive at recruitment

Exclusion Criteria:

* Previous history of bacteriologically confirmed meningococcal disease
* History of clinically significant allergic sensitivity to any vaccine received in the past
* Immunodeficiency
* Any other acute or chronic systemic illness or dependence or abuse of drugs or alcohol
* Language difficulties sufficient to preclude adequate comprehension of the study information
* Possibility of pregnancy
* Receipt of any other vaccine in the previous 4 weeks
* Receipt of any group B vaccine in the past
* Current participation in any other clinical trial
* Generalized acute systemic illness and/or temp >38C on day of vaccination deferral

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MBBS FRCPath, Principal Investigator — Public Health England

REFERENCES:
- [Result] Findlow J, Taylor S, Aase A, Horton R, Heyderman R, Southern J, Andrews N, Barchha R, Harrison E, Lowe A, Boxer E, Heaton C, Balmer P, Kaczmarski E, Oster P, Gorringe A, Borrow R, Miller E. Comparison and correlation of neisseria meningitidis serogroup B immunologic assay results and human antibody responses following three doses of the Norwegian meningococcal outer membrane vesicle vaccine MenBvac. Infect Immun. 2006 Aug;74(8):4557-65. doi: 10.1128/IAI.00466-06. PMID 16861642